CLINICAL TRIAL: NCT02132078
Title: Long-term Follow-up of Lung Transplant Recipients With Diverticulitis
Brief Title: Epidemiology of Diverticulitis in Lung Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Nocito Antonio, PD Dr.med., University of Zurich
Other Study IDs: LTR_Diverticulitis
Record Dates: First submitted 2014-05-04; First posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Lung Transplant Recipients; Diverticulitis
Keywords: Lung transplant recipients; diverticulitis; immunosuppression
MeSH Terms: conditions — Diverticulitis

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Lung transplant recipients with uncomplicated diverticulitis: Retrospective data analysis of treatment, outcome and recurrency-rate
- Lung transplant recipients with complicated diverticulitis: Retrospective data analysis of treatment, outcome and recurrency-rate

SUMMARY:
The purpose of this study is to assess incidence, treatment modalities and outcome of complicated and uncomplicated diverticulitis in highly immunosuppressed lung transplant recipients (LTRs) in order to establish improved treatment strategies in this high risk patient collective.

DETAILED DESCRIPTION:
Sigmoid diverticulitis is common and potentially problematic in immunosuppressed patients. The choice between conservative and surgical treatment for uncomplicated diverticulitis remains unclear, as well as the value of the Hartmann's procedure (HP) for complicated diverticulitis.

Our aim is to assess incidence, treatment options and outcome of complicated and uncomplicated diverticulitis in highly immunosuppressed lung transplant recipients (LTRs) by retrospectively analysing our prospective database of around 400 lung transplant recipients transplanted between 1992 and 2013.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplant recipient
* Diverticulitis

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We want to retrospectively analyse our prospective database of lung transplant recipients at our institution between 1992 and 2013 with diverticulitis episodes.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 1992-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Epidemiology of Diverticulitis in Lung Transplant Recipients | January 1992- December 2013 (22 years)
  Our aim is to assess incidence, treatment options and outcome of complicated and uncomplicated diverticulitis in highly immunosuppressed lung transplant recipients (LTRs) by retrospectively analysing a prospective database of around 400 LTRs transplanted between 1992 and 2013.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Visceral- and Transplant Surgery, University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland